CLINICAL TRIAL: NCT00529984
Title: A Phase I/II Study of Active Immunotherapy With CEA(6D)VRP Vaccine(AVX701)in Patients With Advanced or Metastatic Malignancies Expressing CEA or Stage III Colon Cancer
Brief Title: A Phase I/II Study With CEA(6D) VRP Vaccine in Patients With Advanced or Metastatic CEA-Expressing Malignancies
Acronym: CEA(6D)VRP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AlphaVax, Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVX701; P01CA078673-04 (NIH)
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Colorectal Cancer; Breast Cancer; Lung Cancer; Pancreatic Cancer; Colon Cancer
Keywords: CEA; CEA-expressing malignancies; Metastatic malignancies; VRP Vaccine; Alphavirus replicons; Molecular therapeutics; Stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental)
  Interventions: Biological: AVX701
- Cohort 2 (Experimental)
  Interventions: Biological: AVX701
- Cohort 3 (Experimental)
  Interventions: Biological: AVX701
- Cohort 4 (Experimental)
  Interventions: Biological: AVX701
- Cohort 5 (Experimental)
  Interventions: Biological: AVX701

INTERVENTIONS:
Biological: AVX701 — 4 doses of AVX701 at 4e7 IU given at T=0, 3, 6, 9 weeks. Option for subjects to receive additional immunizations every 3 months after the 4th immunization if no dose-limiting toxicities or is without progressive disease
  Arms: Cohort 1
Biological: AVX701 — 4 doses of AVX701 at 1e8 IU given at T=0, 3, 6, 9 weeks. Option for subjects to receive additional immunizations every 3 months after the 4th immunization if no dose-limiting toxicities or is without progressive disease
  Arms: Cohort 2
Biological: AVX701 — 4 doses of AVX701 at 4e8 IU given at T=0, 3, 6, 9 weeks. Option for subjects to receive additional immunizations every 3 months after the 4th immunization if no dose-limiting toxicities or is without progressive disease
  Arms: Cohort 3
Biological: AVX701 — 4 doses of AVX701 given at the maximally tolerated dose at T=0, 3, 6, 9 weeks. Option for subjects to receive additional immunizations every 3 months after the 4th immunization if no dose-limiting toxicities or is without progressive disease
  Arms: Cohort 4
Biological: AVX701 — 4 Doses of AVX701 given to Stage III colon cancer subjects at the maximally tolerated dose at T=0, 3, 6, 9 weeks. There will be no option for subjects to receive additional immunizations.
  Arms: Cohort 5

SUMMARY:
STUDY OBJECTIVES

1. The primary objective of this protocol is to determine the safety of immunization with CEA(6D) VRP in patients with advanced or metastatic CEA expressing malignancies.
2. The secondary objectives are to evaluate CEA-specific immune response to the immunizations and obtain preliminary data on response rate.

DETAILED DESCRIPTION:
CEA represents an attractive target antigen for immunotherapy since it is over expressed in nearly all colorectal cancers and pancreatic cancers, and is also expressed by some lung and breast cancers, and uncommon tumors such as medullary thyroid cancer, but is not expressed in other cells of the body except for low-level expression in gastrointestinal epithelium [1]. That CEA is a potential target for T cell mediated immune responses in humans is demonstrated by the observation that CEA contains epitopes that may be recognized in an MHC restricted fashion by T cells [2-11]. Specifically, there is support for the existence of human cytolytic T cells (CTLs) that recognize CEA epitopes that bind to MHC molecules HLA- A2, A3, and A24. For the most part, these T cells have been generated by in vitro cultures using antigen-presenting cells pulsed with the epitope of interest to stimulate peripheral blood mononuclear cells. In addition, T cell lines have been generated after stimulation with CEA latex beads, CEA protein-pulsed plastic adherent peripheral blood mononuclear cells, or DCs sensitized with CEA RNA. T cells have also been generated from patients immunized with a vaccinia vector encoding CEA immunogen (discussed below). Using high-performance liquid chromatography mass-spectrometry-based approaches, HLA A2-presented peptides from CEA have been identified in primary gastrointestinal tumors [12]. Of the HLA A2 restricted epitopes of CEA, CAP-1, a nine amino acid sequence, has been shown to stimulate CTLs from cancer patients immunized with vaccinia-CEA. Cap-1(6D) is a peptide analog of CAP-1. Its sequence includes a heteroclitic (nonanchor position) mutation, resulting in an amino acid change from Asn to Asp, to enhance recognition by the T-cell receptor without any change in binding to HLA A2. Compared with the non mutated CAP-1 epitope, Cap-1(6D) has been shown to enhance the sensitization of CTLs by 100 to 1,000 times [3, 5, 13]. CTL lines could be elicited from peripheral blood mononuclear cells of healthy volunteers by in vitro sensitization to the Cap-1(6D) peptide but not to the CAP-1 peptide. These cell lines can lyse human tumor cells expressing endogenous CEA.

ELIGIBILITY:
Inclusion Criteria:

Cohorts 1-4 only:

* Histologically confirmed diagnosis of metastatic malignancy due to a tumor expressing CEA.
* The tumor must express CEA as defined by immunohistochemical staining, CEA blood level, or a tumor known to be universally CEA positive.
* Must have received treatment with standard therapy having a possible overall survival benefit or refused such therapy.
* Must have received and progressed through at least one line of palliative chemotherapy for colorectal, breast, lung, or pancreatic cancer. For other malignancies, if a first line therapy with survival or palliative benefit exists, it should have been administered and there should have been progressive disease.

Cohort 5 Only:

* Histologically confirmed colon cancer (rectal cancer excluded). Since colon cancer is nearly universally CEA positive, CEA staining is not required.
* Documented stage III colon cancer with no evidence of disease.
* One to six months following standard post-operative adjuvant treatment, which should have consisted of 5-fluorouracil and folinic acid or capecitabine with or without oxaliplatin for 4-6 months)

All Cohorts:

* Karnofsky performance status ≥ 70%.
* Estimated life expectancy > 6 months and not expected to require further systemic chemotherapy for at least 3 months.
* Age ≥ 18 years.
* Adequate hematologic function (WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL, and platelets ≥ 100,000/microliter).
* Adequate renal and hepatic function, (serum creatinine < 1.5 mg/dL, bilirubin ≤ 1.5 mg/dL, and ALT and AST ≤ 2.5 x upper limit of normal).
* Patients who have received CEA-targeted immunotherapy, if treatment was discontinued at least 3 months before enrollment.
* Patients who are taking medications that do not have a known history of immunosuppression are eligible for this trial.
* Ability to understand and provide signed informed consent.
* Ability to return to Duke University Medical Center for adequate follow-up, as required by protocol.

Exclusion Criteria:

* Concurrent cytotoxic chemotherapy or radiation therapy (must be at least 3 months between any prior CEA-targeted immunotherapy and study treatment and at least 4 weeks between any other prior therapy and study treatment).
* Patients with previously resected brain metastases will be permitted if a CT or MRI scan shows no metastasis within 1 month before enrollment.
* History of autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
determine the safety of immunization with CEA(6D) VRP | 2.5 years

SECONDARY OUTCOMES:
evaluate CEA-specific immune response to immunizations | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morse, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States